CLINICAL TRIAL: NCT00739505
Title: A Multicenter, Open-Label, Dose Escalating Study of the Safety, Tolerability and Pharmacology of Human Recombinant Tissue Non-Specific Alkaline Phosphatase Fusion Protein Asfotase Alfa in Adults With Hypophosphatasia (HPP)
Brief Title: Safety Study of Human Recombinant Tissue Non-Specific Alkaline Phosphatase Fusion Protein Asfotase Alfa in Adults With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENB-001-08
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia (HPP)
Keywords: Hypophosphatasia; Bone Disease; Soft Bones; Low Alkaline Phosphatase; genetic metabolic disorder; alkaline phosphatase; tissue non-specific alkaline phosphatase; rickets; osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia | interventions — asfotase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): 3 HPP patients are to be enrolled in Cohort 1 and receive a single IV dose and three weekly SC doses of Asfotase Alfa . End of Study for patients in Cohort 1 is at 8 weeks.
  Interventions: Biological: Asfotase Alfa
- Cohort 2 (Experimental): Cohort 2 will begin when the safety and PK data for Cohort 1 weeks 1-4 has been reviewed by the DSMB. Cohort 2 will enroll 3 HPP patients and will receive a higher dose level than Cohort 1. Cohort 2 patients will have a single IV dose and three weekly SC doses of Asfotase Alfa . End of Study for patients in Cohort 2 is at 8 weeks.
  Interventions: Biological: Asfotase Alfa

INTERVENTIONS:
Biological: Asfotase Alfa — The initial IV dose to be administered to patients was set at one-tenth the no adverse effect level (NOAEL) as determined by one month toxicology studies in animals in which Asfotase Alfa was administered as a single weekly IV dose. The SC doses to be administered are lower than the IV doses and are thought to be near or at the anticipated daily efficacious dose. Dosing will be as follows:
  Cohort 1: In Week 1, patients will receive an IV infusion of Asfotase Alfa at a dose of 3 mg/kg. In Weeks 2, 3 and 4, patients will receive weekly SC injections of Asfotase Alfa at a dose of 1 mg/kg SC.
  Arms: Cohort 1
Biological: Asfotase Alfa — Cohort 2: In Week 1, patients will receive an IV infusion of Asfotase Alfa at a dose of 7 mg/kg. In Weeks 2, 3 and 4, patients will receive weekly SC injections of Asfotase Alfa at a dose of 1.5 mg/kg SC.
  Arms: Cohort 2

SUMMARY:
This clinical trial studies the safety, tolerability, and pharmacology of asfotase alfa when given to adults with HPP.

DETAILED DESCRIPTION:
Asfotase alfa was formerly referred to as ENB-0040

Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are no approved disease-modifying treatments for patients with this disease. There is also limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

ELIGIBILITY:
Inclusion Criteria:

In order to qualify for participation, patients must meet all of the following criteria:

* Patients must provide written informed consent, including privacy authorization, prior to participation.
* Women of childbearing potential must sign the Women of Childbearing Potential Addendum and must be using an acceptable method of birth control. Women considered not of childbearing potential must be surgically sterile (total hysterectomy, bilateral salpingo-oophorectomy, or tubal ligation) or post-menopausal, which is defined as a complete cessation of menstruation for at least one year after the age of 45 years. All women must have a serum pregnancy test conducted at Screening prior to enrollment and the results must be negative.
* Be between 18 and 80 years of age at the time of consent
* Patients must be medically stable in the opinion of the Investigator.
* Patients must be willing to comply with study procedures and the visit schedule.
* Pre-established clinical diagnosis of HPP as indicated by:

  * a. Serum alkaline phosphatase at least 3 SD below the mean for age
  * b. Radiologic evidence of osteopenia or osteomalacia
  * c. Two or more HPP-related findings:

    * i. Plasma pyridoxal 5'-phosphate at least 2.5 SD above the mean (no vitamin B6 administered for at least 1 week prior to determination
    * ii. History of rickets
    * iii. History of premature loss of deciduous teeth
    * iv. Bone deformity consistent with osteomalacia or past history of rickets
    * v. History of any one of the following:

      * 1. Non-traumatic fracture
      * 2. Pseudofracture
      * 3. Non-healing fracture

Exclusion Criteria:

In order to qualify for participation, patients must not meet any of the following criteria:

* Women who are pregnant or lactating.
* History of sensitivity to any of the constituents of the study drug.
* Low levels of serum calcium, magnesium or phosphate.
* Serum 25(OH) vitamin D level below 9.2 ng/mL.
* Elevated serum creatinine or parathyroid hormone level.
* Known cause of hypophosphatasemia other than HPP.
* Current or prior clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal condition and/or other major disease which, in the opinion of the investigator, precludes study participation.
* Treatment with a bisphosphonate or parathyroid hormone (PTH) within 6 months prior to the start of Asfotase Alfa administration.
* Participation in an interventional or investigational drug study within 30 days prior to study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of Asfotase Alfa given intravenously and given subcutaneously. | Within the first 2 months (8 weeks).

SECONDARY OUTCOMES:
To assess the pharmacokinetics (PK) of Asfotase Alfa given intravenously and subcutaneously | Within the first 2 months (8 weeks)
To assess the bioavailability of the subcutaneous Asfotase Alfa | Within the first 2 months (8 weeks)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Barnes Jewish Hospital- Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
- Department of Pediatrics & Child Health, Health Sciences Centre Winnipeg, University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Millan JL, Narisawa S, Lemire I, Loisel TP, Boileau G, Leonard P, Gramatikova S, Terkeltaub R, Camacho NP, McKee MD, Crine P, Whyte MP. Enzyme replacement therapy for murine hypophosphatasia. J Bone Miner Res. 2008 Jun;23(6):777-87. doi: 10.1359/jbmr.071213. PMID 18086009
- [Background] Drake MT, Khosla S. Bone-targeted replacement therapy for hypophosphatasia. J Bone Miner Res. 2008 Jun;23(6):775-6. doi: 10.1359/jbmr.080305. No abstract available. PMID 18318644
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Healthcare Providers — http://www.hypophosphatasia.com/hcp/
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org